CLINICAL TRIAL: NCT05511818
Title: Radicle™ Rest: A Randomized, Blinded, Placebo-controlled, Direct-to-consumer Study Assessing the Impact of Plant Derived Cannabinoids on Sleep and Overall Health Outcomes
Brief Title: Radicle Rest: A Study of Cannabinoids on Sleep and Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-22D03
Record Dates: First submitted 2022-08-10; First posted 2022-08-23 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Sleep; Sleep Disturbance; Sleep Disorder
MeSH Terms: conditions — Parasomnias; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender at birth then randomized to one of the study arms
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Placebo Control 1 (Placebo Comparator): Rest Product Form 1 - control
  Interventions: Dietary Supplement: Rest Study Product Usage
- Placebo Control 2 (Placebo Comparator): Rest Product Form 2 - control
  Interventions: Dietary Supplement: Rest Study Product Usage
- Placebo Control 3 (Placebo Comparator): Rest Product Form 3 - control
  Interventions: Dietary Supplement: Rest Study Product Usage
- Active Product 1.1 (Experimental): Rest Product Form 1 - active product 1
  Interventions: Dietary Supplement: Rest Study Product Usage
- Active Product 1.2 (Experimental): Rest Product Form 1 - active product 2
  Interventions: Dietary Supplement: Rest Study Product Usage
- Active Product 1.3 (Experimental): Rest Product Form 1 - active product 3
  Interventions: Dietary Supplement: Rest Study Product Usage
- Active Product 1.4 (Experimental): Rest Product Form 1 - active product 4
  Interventions: Dietary Supplement: Rest Study Product Usage
- Active Product 2.1 (Experimental): Rest Product Form 2 - active product 1
  Interventions: Dietary Supplement: Rest Study Product Usage
- Active Product 2.2 (Experimental): Rest Product Form 2 - active product 2
  Interventions: Dietary Supplement: Rest Study Product Usage
- Active Product 3.1 (Experimental): Rest Product Form 3 - active product 1
  Interventions: Dietary Supplement: Rest Study Product Usage
- Active Product 3.2 (Experimental): Rest Product Form 3 - active product 2
  Interventions: Dietary Supplement: Rest Study Product Usage
- Placebo Control 4 (Placebo Comparator): Rest Product Form 4 - control
  Interventions: Dietary Supplement: Rest Study Product Usage
- Active Product 4 (Experimental): Rest Product Form 4 - active product 1
  Interventions: Dietary Supplement: Rest Study Product Usage

INTERVENTIONS:
Dietary Supplement: Rest Study Product Usage — Participants will use their Radicle Rest study product as directed for a period of 4 weeks.

SUMMARY:
A randomized, blinded, placebo-controlled, direct-to-consumer study assessing the impact of plant derived cannabinoids on sleep and overall health outcomes

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled study conducted with up to 300 adult participants per study arm, age 21 and older and residing in the United States.

Eligible participants will (1) endorse a desire for better sleep, (2) indicate a willingness to refrain from taking cannabinoids during the study period, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants with known liver disease, heavy drinkers, and those who are pregnant, trying to become pregnant, or breastfeeding will be excluded. Those taking medications that warn against grapefruit consumption will be excluded.

Self-reported data are collected electronically from eligible participants over 5 weeks. Participant reports of health indicators will be collected during baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and older
* Resides in the United States
* Endorses a desire for better sleep
* Selects sleep as a primary reason for taking a cannabinoid product
* Expresses a willingness to refrain from taking any non-study cannabinoid product (i.e. CBD, CBG, CBC, CBN, THC) for the duration of participant engagement (5 weeks)
* Expresses an interest in taking a study product and not knowing the product identity until the end of the study

Exclusion Criteria:

* Pregnant, trying to become pregnant, or breastfeeding
* Reports a diagnosis of liver disease
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Lack of reliable daily access to the internet
* Reports taking any medication that warns against grapefruit consumption

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2679 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Change in sleep disturbance | 4 weeks
  Mean difference in sleep disturbance score as assessed by Patient Reported Outcome Measurement System (PROMIS) Sleep Disturbance Short Form 8A (scale 8-40; where higher scores correspond to greater sleep disturbance)

SECONDARY OUTCOMES:
Change in overall well-being | 4 weeks
  Mean difference in well-being score as assessed by World Health Organization 5 (WHO 5; scale 0-25; with 0 representing the worst imaginable well-being and 25 representing the best imaginable well-being)
Change in overall quality of life (QOL) | 4 weeks
  Mean difference in QOL score as assessed by Kemp QOL (scale 1-7; with 1 representing very poor QOL and 7 representing excellent QOL)
Change in anxiety | 4 weeks
  Mean difference in anxiety score as assessed by PROMIS Anxiety 4A (scale 4-20; with higher scores corresponding to more severe anxiety)
Change in pain | 4 weeks
  Mean difference in pain score as assessed by the Pain on average, Enjoyment of life, and General activity score (PEG; scale 0-10; with 0 representing no pain and 10 representing the worst pain imaginable that completely interferes with enjoyment of life and general activities)
Change in stress | 4 weeks
  Mean difference in stress score as assessed by PROMIS Stress 4A (scale 4-20; where higher scores correspond to more severe stress)
Change in fatigue | 4 weeks
  Mean difference in fatigue score as assessed by PROMIS Fatigue 4A (scale 4-20; where higher scores correspond to more severe fatigue)
Minimal clinically important difference (MCID) in sleep disturbance | 4 weeks
  Likelihood of achieving a MCID in sleep disturbance, as measured by PROMIS Sleep Disturbance Short Form 8A (scale 8-40; where higher scores correspond to greater sleep disturbance)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com